CLINICAL TRIAL: NCT05202041
Title: Diagnostic Performance and Prognostic Ability of AccuFFRangio for Non-IRA in NSTE-ACS Patients
Brief Title: Non-IRA Functional Evaluation With AccuFFRangio in NSTE-ACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFCA20211130
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Non ST Segment Elevation Acute Coronary Syndrome; Coronary Artery Disease; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AccuFFRangio Group (Experimental): NSTE-ACS patients with multiple lesions who met the requirements of the study were enrolled and received coronary angiography. First, the revascularization of the criminal vessel (PCI) was completed. The patients were randomly grouped and divided into AccuFFRangio Group and Angiography Group if the treatment results were good. The AccuFFRangio Group was defined as non-IRA of these patients who were treated with PCI after angio-FFR measurement with FFR≤0.8.
  Interventions: Other: AccuFFRangio-guided strategy
- Angiography Group (Active Comparator): The Angiography Group was defined as PCI treatment for non-IRA when diameter stenosis > 70% based on angiographic results.
  Interventions: Other: Angiography-guided strategy

INTERVENTIONS:
Other: AccuFFRangio-guided strategy — In this study, the AccuFFRangio-guided strategy will be applied to in the AccuFFRangio group in which calculation of the AccuFFRangio values of all target coronary arteries with lesions with diameter stenosis of ≥ 50% (visual estimation) and with suitability to PCI revascularization will be carried out. If AccuFFRangio ≤ 0.80, then simultaneous PCI revascularization of target blood vessels will be carried out. If AccuFFRangio > 0.80, then no PCI revascularization of target blood vessels will be carried out.
  Arms: AccuFFRangio Group
Other: Angiography-guided strategy — In this study, CAG-guided strategy will be used for the control group, i.e., in accordance with current guideline recommendations, all target coronary arteries with lesions with diameter stenosis of ≥ 70% (visual estimation) and suited for PCI revascularization will undergo PCI revascularization.
  Arms: Angiography Group

SUMMARY:
This is a prospective, single-center clinical trial. AccuFFRangio (ArteryFlow Technology Co., Ltd., Hangzhou, China) is a novel method for evaluating the functional significance of coronary stenosis by computing the pressure in the vessel based on angiographic images. The purpose of this study is to investigate the diagnostic performance and prognostic ability of AccuFFRangio for non-IRA in NSTE-ACS patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* Non-ST-segment elevation acute coronary syndrome patients with at least 1 non-IRA
* Diameter stenosis of 50%-90% by visual estimate
* Reference vessel size > 2 mm in stenotic segment by visual estimate

Exclusion Criteria:

* LVEF ≤ 40%
* eGFR < 60 mL/min
* Allergy to contrast media, adenosine
* Prior CABG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-02-15 (Estimated); Primary Completion 2023-02-14 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Vessel-oriented composite endpoints (VOCEs) | 1 year
  Composite of vessel-related cardiovascular death, vessel-related myocardial infarction, and ischemia-driven target vessel revascularization.
Post-PCI AccuFFRangio | 1 year
  AccuFFRangio limits to yield no VOCEs.

SECONDARY OUTCOMES:
Cost analysis | 1 year
  Cost savings of AccuFFRangio-guided strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Song, MD, Study Chair — Wuhan Aisa Heart Hospital

IPD SHARING:
Plan to Share IPD: No